CLINICAL TRIAL: NCT07299786
Title: Multicomponent Exercise Prescription Through Telerehabilitation for Older Adults With Multiple Chronic Conditions in Antioquia, Colombia
Brief Title: Telerehabilitation With Multicomponent Exercise for Older Adults With Multiple Chronic Conditions
Acronym: TELEREAHB-COL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Universitaria Maria Cano (Other)
Collaborators: Universidad Iberoamericana A.C., Mexico (Other)
Responsible Party: Principal Investigator, Silvia Patricia Betancur Bedoya, Principal Investigator, Fundacion Universitaria Maria Cano
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 013008001-2024311
Record Dates: First submitted 2025-11-28; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Multiple Comorbidity
Keywords: telerehabilitation; Multicomponent Exercise; Multiple Chronic Conditions
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: This study follows a parallel-group design with two intervention arms: a Telerehabilitation Group (TRG) and a Conventional Home-Based Physiotherapy Group (HBG). Participants will be randomly assigned in a 1:1 ratio, stratified by primary diagnosis and sex, to ensure balanced distribution between groups. Each participant will remain in the same group throughout the 12-week intervention period.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study was conducted as a single-blind trial. Both participants and outcome assessors were blinded to group allocation. Participants were informed that they would take part in one of two exercise-based physiotherapy programs, without being told which one was the experimental (telerehabilitation) or the control (home-based physiotherapy) intervention. Outcome assessors responsible for pre- and post-intervention evaluations were also blinded to participant allocation to minimize assessment bias. The physiotherapists who delivered the interventions were not blinded due to the nature of the procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (TRG) (Experimental): Participants in the Telerehabilitation Group (TRG) will take part in a 12-week multicomponent exercise program delivered online through Microsoft Teams. Sessions will be held twice per week, lasting 45 minutes each, and will include aerobic, strength, flexibility, and balance exercises. Intensity will be individually adjusted according to perceived exertion and functional status. A physiotherapist will conduct the sessions in real time, providing continuous supervision, feedback, and safety monitoring.
  Interventions: Behavioral: Multicomponent Exercise via Telerehabilitation
- Home-Based Physiotherapy Group (HBG) (Active Comparator): Participants in the Home-Based Physiotherapy Group (HBG) received a 12-week in-home physiotherapy program conducted by a physiotherapist who visited the participants' homes twice per week. Each session lasted approximately 45 minutes and included aerobic, strength, flexibility, and balance exercises, following the same structure as the telerehabilitation protocol. The exercises were individualized according to the participant's clinical condition and physical capacity. Progress and safety were monitored directly during each home session.
  Interventions: Behavioral: Home-Based Physiotherapy

INTERVENTIONS:
Behavioral: Multicomponent Exercise via Telerehabilitation — A supervised multicomponent exercise program delivered remotely through Microsoft Teams. The program includes aerobic, strength, flexibility, and balance exercises performed twice per week for 12 weeks, under real-time supervision by a physiotherapist. The exercises are individualized according to each participant's health status and physical capacity.
  Other Names: TRG
  Arms: Telerehabilitation Group (TRG)
Behavioral: Home-Based Physiotherapy — A physiotherapist-led multicomponent exercise program conducted in person at the participant's home. The intervention includes aerobic, strength, flexibility, and balance exercises, delivered twice per week for 12 weeks. The physiotherapist provides individualized progression, monitors adherence, and ensures participant safety during each home session.
  Other Names: HBG
  Arms: Home-Based Physiotherapy Group (HBG)

SUMMARY:
The goal of this clinical trial is to learn if a multicomponent exercise program delivered through telerehabilitation improves physical fitness and quality of life in older adults with multiple chronic conditions living in Antioquia, Colombia.

The main questions it aims to answer are:

Does telerehabilitation with multicomponent exercise improve physical performance compared to home-based physiotherapy provided in person by a physiotherapist?

Does this program enhance participants' quality of life and functional independence?

Participants will:

Join a 12-week exercise program with two 45-minute online sessions per week, led by a physiotherapist through Microsoft Teams.

Perform exercises including aerobic, strength, flexibility, and balance training, adapted to their health condition.

Complete pre- and post-intervention assessments of physical function (Senior Fitness Test, SPPB) and quality of life (WHOQOL-BREF).

Researchers will compare the telerehabilitation group to a home-based physiotherapy group, in which physiotherapists visit participants at their homes, to determine whether the online multicomponent exercise intervention is effective, safe, and feasible for older adults with multiple chronic conditions.

DETAILED DESCRIPTION:
This study is a randomized, single-blind, parallel-group controlled clinical trial designed to evaluate the implementation and effects of a multicomponent exercise program delivered through synchronous telerehabilitation in older adults with multiple chronic conditions living in Antioquia, Colombia.

Population aging has led to a growing prevalence of multimorbidity, characterized by the coexistence of cardiovascular, respiratory, metabolic, and musculoskeletal conditions. This clinical complexity is commonly associated with declines in physical function, increased frailty, loss of independence, and reduced quality of life. Although exercise-based rehabilitation is a key component of chronic disease management, access to supervised programs remains limited for many older adults due to geographic barriers, mobility restrictions, and resource constraints, particularly in low- and middle-income settings.

Telerehabilitation, defined as the remote delivery of rehabilitation services through information and communication technologies, has emerged as an alternative approach to improve access to physiotherapy services while maintaining professional supervision. Multicomponent exercise programs that integrate aerobic, resistance, flexibility, and balance training have demonstrated benefits for physical and functional health in older populations. However, there is limited evidence regarding the use of supervised telerehabilitation models for older adults with multimorbidity in Colombia.

Participants are allocated in a 1:1 ratio to either a Telerehabilitation Group or a Home-Based Physiotherapy Group. Randomization is stratified by sex and primary diagnosis to promote balance between groups. Outcome assessors are blinded to group allocation.

The telerehabilitation intervention consists of a structured, supervised multicomponent exercise program delivered in real time using videoconferencing technology. Sessions are conducted twice weekly over a 12-week period and follow a standardized format that includes warm-up activities, aerobic conditioning, resistance exercises using body weight or elastic bands, flexibility training, balance exercises, and cool-down. Exercise intensity and progression are individualized based on functional capacity, health status, and participant tolerance. All sessions are supervised synchronously by a licensed physiotherapist, who provides guidance, monitors responses to exercise, and applies predefined safety procedures.

The comparison group receives an equivalent multicomponent exercise program delivered face-to-face in the participant's home by a physiotherapist over the same intervention period. Session structure, exercise components, and progression principles are comparable between groups, with the primary difference being the mode of delivery. Both groups receive standardized educational guidance related to physical activity, healthy aging, and self-management strategies.

Assessments are conducted at baseline and immediately after completion of the intervention period. Study procedures include monitoring adherence, documenting attendance, and recording any adverse events occurring during supervised exercise sessions. These elements are used to evaluate feasibility, acceptability, and safety of the intervention in both delivery modalities.

Ethical approval was obtained from the Research Ethics Committee of Fundación Universitaria María Cano. All participants provided written informed consent prior to enrollment. Participant confidentiality and data protection are ensured in accordance with institutional protocols and national regulations, including secure management of digital platforms used for telerehabilitation.

This trial aims to generate context-specific evidence on the use of supervised telerehabilitation as a strategy to deliver physiotherapy services to older adults with multiple chronic conditions, supporting future integration of digital rehabilitation models into clinical practice and public health initiatives in Colombia.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years or older.
* Diagnosed with a chronic cardiorespiratory condition (e.g., chronic obstructive pulmonary disease, asthma, heart failure, or ischemic heart disease).
* May present other stable chronic comorbidities (e.g., metabolic or musculoskeletal diseases).
* Medically stable and cleared by a physician to participate in moderate exercise.
* Able to stand and walk independently, with or without assistive devices.
* Have access to a device with an internet connection (computer, tablet, or smartphone) for online sessions.
* Cognitive ability to follow instructions and communicate with the physiotherapist.
* Willingness to provide informed consent and comply with the study procedures.

Exclusion Criteria:

* Severe dementia or cognitive impairment preventing participation.
* Uncontrolled epilepsy or recent seizure history.
* Recent major surgery (within the past 3 months).
* Delirium or acute confusional state.
* Recent acute myocardial infarction or unstable angina.
* Uncontrolled arrhythmias. -Dissecting aortic aneurysm.-
* Severe aortic stenosis.
* Acute endocarditis or pericarditis.
* Uncontrolled hypertension. -Acute thromboembolic disease.- Any medical condition or instability that, in the investigator's judgment, would make participation unsafe or inappropriate.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Change in Physical Performance Measured by the Short Physical Performance Battery (SPPB) | Baseline and 12 weeks post-intervention
  The Short Physical Performance Battery (SPPB) is a standardized test that assesses lower extremity function through three components: balance, gait speed, and chair stand performance. Each component is scored from 0 to 4, with a total score ranging from 0 to 12, where higher scores indicate better physical performance. The SPPB has been validated as a predictor of functional capacity, frailty, and disability in older adults. In this study, the SPPB will be used to evaluate changes in physical performance before and after the 12-week intervention in both groups.
Change in Physical Fitness Measured by the Senior Fitness Test (SFT) | Baseline and 12 weeks post-intervention
  The Senior Fitness Test (SFT) is a standardized battery designed to assess physical fitness in older adults across multiple components of functional capacity. It includes six subtests evaluating lower-body strength, upper-body strength, aerobic endurance, flexibility, agility, and dynamic balance: chair stand, arm curl, 2-minute step, chair sit-and-reach, back scratch, and 8-foot up-and-go.
  Each subtest is scored independently using performance-based measures. There is no single composite score for the SFT. The minimum and maximum values for each subtest are as follows:
  Chair Stand Test: number of repetitions completed in 30 seconds (minimum = 0 repetitions; no fixed maximum).
  Arm Curl Test: number of repetitions completed in 30 seconds (minimum = 0 repetitions; no fixed maximum).
  2-Minute Step Test: number of steps completed in 2 minutes (minimum = 0 steps; no fixed maximum).
  Chair Sit-and-Reach Test: distance reached in centimeters relative to the toes (negative values indicate

SECONDARY OUTCOMES:
Change in Quality of Life Measured by the WHOQOL-BREF Questionnaire | Baseline and 12 weeks post-interventio
  The World Health Organization Quality of Life Instrument (WHOQOL-BREF) is a validated questionnaire that assesses quality of life across four domains: physical health, psychological health, social relationships, and environment. The instrument consists of 26 items rated on a 5-point Likert scale. Domain scores are calculated and transformed to a 0-100 scale following World Health Organization guidelines.
  For all domains and the overall quality of life score, higher scores indicate better perceived quality of life, while lower scores indicate poorer perceived quality of life.
  In this study, the WHOQOL-BREF will be administered at baseline and after the 12-week intervention to evaluate changes in overall and domain-specific quality of life in both study groups.

OTHER OUTCOMES:
Participant Satisfaction with the Telerehabilitation Program | At the end of the 12-week intervention
  Participant satisfaction will be assessed through a structured questionnaire designed to evaluate perceptions of the telerehabilitation experience, including ease of use, communication with the physiotherapist, perceived benefits, session duration, and overall satisfaction. Responses will be rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree), with higher scores indicating greater satisfaction. Open-ended questions will allow qualitative feedback on the strengths and limitations of the program.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Universitaria María Cano, Envigado, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional and ethical restrictions. Only aggregated and anonymized data will be published in scientific reports and peer-reviewed journals.